CLINICAL TRIAL: NCT03530501
Title: Effects of Very-low Ketogenic Diet in Gut Microbiota and Its Restitution With the Use of Synbiotic Supplementation in Patients Following a Weight Loss Programme (Pronokal Method)
Brief Title: Effect of Very-low Calorie Diet and Synbiotic Supplementation in Gut Microbiota (Pronokal Method)
Acronym: Pronokal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JGA-BIOPNK-2016-01
Record Dates: First submitted 2018-04-05; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-04

CONDITIONS: Weight Loss; Inflammation
Keywords: microbiota; obesity
MeSH Terms: conditions — Weight Loss; Inflammation; Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Very low calorie ketogenic diet followed by low calorie diet
  Interventions: Other: Diet
- Synbiotic1+synbiotic2 (Experimental): Very low calorie ketogenic diet supplemented with synbiotic 1 followed by low calorie diet supplemented with synbiotic2
  Interventions: Other: Diet; Dietary Supplement: Synbiotic1; Dietary Supplement: Synbiotic2
- placebo +synbiotic2 (Experimental): Very low calorie ketogenic diet supplemented with placebo followed by low calorie diet supplemented with synbiotic2
  Interventions: Other: Diet; Dietary Supplement: Synbiotic2

INTERVENTIONS:
Other: Diet — Very low calorie ketogenic diet followed by low calorie diet
Dietary Supplement: Synbiotic1 — B. lactis, Lactobacillus rhamnosus, B. longum ES1 and prebiotics fiber
  Arms: Synbiotic1+synbiotic2
Dietary Supplement: Synbiotic2 — B. animalis subsp. lactis and prebiotics fiber
  Arms: Synbiotic1+synbiotic2; placebo +synbiotic2

SUMMARY:
The present study aimed to investigate the changes produced in gut microbiota by a very-low-calorie-ketogenic diet followed by a low calorie diet, whether the use of synbiotics is able to modulate gut microbiota diversity and composition and its association with gut permeability and inflammation

DETAILED DESCRIPTION:
All participants followed a very-low-calorie ketogenic diet according to a commercial weight loss program (Pronokal method), which includes lifestyle and behavioural modification support. This method is based on high-biological-value protein preparations which contained 15 g protein, 4 g carbohydrates, 3 g fat and 50 mg docosahexaenoic acid, and provided 90-110 kcal. The study was divided in two phases. The first phase consists of a very-low-calorie ketogenic diet (600-800 kcal/day), low in carbohydrates and lipids. Throughout this ketogenic phase, supplements of vitamins and minerals such as K, Na, Mg, Ca and omega-3 fatty acids were provided. In this study the ketogenic step was maintained for 2 months. Then, the patients started a low-calorie diet (800-1500 kcal/day) which lasted two months.

During the first phase consisting of a very-low-calorie ketogenic diet, subjects were randomly divided into two groups, the treatment group who received synbiotic supplementation as capsules, a complex of B. lactis, Lactobacillus rhamnosus, B. longum ES1 and prebiotics fiber (synbiotic 1) and the control group who received a placebo. During the second phase consisting of a low-calorie diet, the treatment group received synbiotic supplementation as capsules consisting of B. animalis subsp. lactis and prebiotics fiber (synbiotic 2) (synbiotic1 + synbiotic 2 group), while the control group was divided into two groups: one continued receiving a placebo (control group) whilst the other group received synbiotic 2 (placebo + synbiotic2 group).

ELIGIBILITY:
Inclusion Criteria:

* body mass index ≥ 30 kg/m2
* stable body weight in the previous 3 months

Exclusion Criteria:

* Diabetes mellitus
* Obesity induced by endocrine disorders or by drugs
* Gastrointestinal disorders
* Use of antibiotics, probiotic or prebiotic agent which could modify microbiota in the previous 3 months
* Severe depression or any other psychiatric disease
* Abuse of narcotics or alcohol
* Severe hepatic insufficiency
* Any type of renal insufficiency or gout episodes
* Neoplasia
* Previous events of cardiovascular or cerebrovascular disease
* Renal lithiasis
* Uncontrolled hypertension and hydroelectrolytic alterations
* Females with child-bearing potential, who were pregnant, breast-feeding, intending to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Changes produced in the composition and diversity of gut microbiota by the use of synbiotics during a dietary intervention | At baseline and at 4 months
  Fecal samples were collected at baseline and at the end of dietary intervention. Fecal DNA was extracted and Gut microbiota analysis was achieved by using high-throughput sequencing

SECONDARY OUTCOMES:
Changes in intestinal permeability markers produced by the use of synbiotics during a dietary intervention | At baseline and at 4 months
  Blood samples were collected at baseline and at the end of study. Plasma Zonulin levels were measured by enzyme linked immunosorbent assay
Changes in intestinal inflammation markers produced by the use of synbiotics during a dietary intervention | At baseline and at 4 months
  Blood samples were collected at baseline and at the end of study. Plasma C-reactive protein levels were measured by enzyme linked immunosorbent assay
Changes in microbial translocation markers produced by the use of synbiotics during a dietary intervention | At baseline and at 4 months
  Blood samples were collected at baseline and at the end of study. Plasma lipopolysaccharide binding protein levels were measured by enzyme linked immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel García-Almeida, MD, Study Director — Hospital Universitario Virgen de la Victoria
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Spain

REFERENCES:
- [Derived] Gutierrez-Repiso C, Hernandez-Garcia C, Garcia-Almeida JM, Bellido D, Martin-Nunez GM, Sanchez-Alcoholado L, Alcaide-Torres J, Sajoux I, Tinahones FJ, Moreno-Indias I. Effect of Synbiotic Supplementation in a Very-Low-Calorie Ketogenic Diet on Weight Loss Achievement and Gut Microbiota: A Randomized Controlled Pilot Study. Mol Nutr Food Res. 2019 Oct;63(19):e1900167. doi: 10.1002/mnfr.201900167. Epub 2019 Aug 29. PMID 31298466